CLINICAL TRIAL: NCT03172988
Title: Impact of Perioperative Dexamethasone and Flurbiprofen Axetil on Long-term Survival After Surgery for Non-small Cell Lung Cancer: A 2x2 Factorial Randomized Controlled Trial
Brief Title: Dexamethasone, Flurbiprofen Axetil and Long-term Survival After Lung Cancer Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol violation occurred frequently during the postoperative period.
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017[1359]-2
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Surgery; Dexamethasone; Flubiprofen Axetil; Long-term Effects Secondary to Cancer Therapy in Adults
Keywords: Carcinoma, Non-Small-Cell Lung; Surgery; Dexamethasone; Flurbiprofen axetil; Long-term survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dexamethasone; dexamethasone 21-phosphate; Saline Solution; flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexamethasone and flurbiprofen axetil (Experimental): Dexamethasone 10 mg is administered before anesthesia induction. Flurbiprofen axetil 50 mg is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 2 mg/ml flurbiprofen axetil, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Dexamethasone; Drug: Flurbiprofen axetil
- Dexamethasone and lipid microsphere (Experimental): Dexamethasone 10 mg is administered before anesthesia induction. Lipid microsphere 5 ml is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 20 ml lipid microsphere, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Dexamethasone; Drug: Lipid microsphere
- Normal saline and flurbiprofen axetil (Experimental): Normal saline 2 ml is administered before anesthesia induction. Flurbiprofen axetil 50 mg is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 2 mg/ml flurbiprofen axetil, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Normal saline; Drug: Flurbiprofen axetil
- Normal saline and lipid microsphere (Placebo Comparator): Normal saline 2 ml is administered before anesthesia induction. Lipid microsphere 5 ml is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg sufentanil and 20 ml lipid microsphere, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Interventions: Drug: Normal saline; Drug: Lipid microsphere

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10 mg is administered before anesthesia induction.
  Other Names: Dexamethasone sodium phosphate injection
  Arms: Dexamethasone and flurbiprofen axetil; Dexamethasone and lipid microsphere
Drug: Normal saline — Normal saline 2 ml is administered before anesthesia induction.
  Arms: Normal saline and flurbiprofen axetil; Normal saline and lipid microsphere
Drug: Flurbiprofen axetil — Flurbiprofen axetil 50 mg is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 2 mg/ml flurbiprofen axetil, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Other Names: Flurbiprofen axetil injection
  Arms: Dexamethasone and flurbiprofen axetil; Normal saline and flurbiprofen axetil
Drug: Lipid microsphere — Lipid microsphere 5 ml is administered before the start of surgery. Postoperative analgesia is provided with a patient-controlled analgesia pump, which is established with 100 ml of 1.25 μg/ml sufentanil and 20 ml lipid microsphere, programmed to deliver a 2 ml bolus with a lockout interval of 6-8 min and a background infusion of 1 ml/h.
  Other Names: Lipid microsphere injection
  Arms: Dexamethasone and lipid microsphere; Normal saline and lipid microsphere

SUMMARY:
Surgical resection is the first choice treatment for patients with non-small-cell lung cancer. Despite of advances in surgical techniques, the long-term survival rate of postoperative patient is far from optimal. In a recent retrospective cohort study of the applicants, 588 patients after surgery for non-small-cell lung cancer were followed up for a medium of 5.2 years. The results showed that perioperative use of dexamethasone was associated with prolonged survival; perioperative use of flurbiprofen axetil was also associated with a slightly longer survival but not statistically significant. Further analysis showed that combined administration of dexamethasone and flurbiprofen axetil had additive effect in prolonging survival. We hypothesize that, for patients undergoing surgery for non-small-cell lung cancer, perioperative administration of dexamethasone and flurbiprofen axetil may improve long-term survival. However, evidences from randomized controlled trials are still lacking in this aspect.

DETAILED DESCRIPTION:
Surgical resection is the first choice treatment for patients with non-small-cell lung cancer. Although improvements of surgical techniques have reduced the incidence of complications, the long-term survival rate of postoperative patient is far from optimal. Cancer metastasis and recurrence are the main reasons that lead to long-term postoperative death. It is unavoidable that some cancer cells will be disseminated into the blood circulation or the lymphatic systems during surgery. The development of metastasis and recurrence are dependent on the balance between the immune function of the body and the cancer-promoting factors during the perioperative period.

Studies showed that surgical stress inhibits the cytotoxic effects of natural killer cells and the activity of T cells, and thus leads to immunosuppression of the body. Furthermore, perioperative management such as anesthetic techniques, anesthetics and related drugs, blood transfusion and hypothermia can also affect immune function. For example, studies showed that inhalational anesthetics and opioids aggravate immunosuppression, and may lead to worse outcome; whereas regional anesthesia and non-steroid anti-inflammatory drugs relieve immunosuppression, and thus may improve outcome. Glucocorticoids (mainly dexamethasone) are frequently used for prevention of postoperative nausea and vomiting. A recent retrospective study showed that, for patients undergoing surgery for pancreatic cancer, perioperative use of dexamethasone was associated with improved long-term survival. However, prospective randomized controlled trials are still lacking to demonstrate the relationship between perioperative management and long-term outcome in cancer patients.

A recent retrospective cohort study of the applicants recruited 588 patients after surgery for non-small-cell lung cancer and performed a postoperative follow-up for a medium of 5.2 years. After adjusting the confounding factors with multivariate logistic regression model, perioperative use of dexamethasone (medium dose 10 mg, for prevention of postoperative nausea and vomiting) was associated with prolonged survival (HR 0.70, 95% CI 0.54-0.89; P = 0.004); perioperative use of flurbiprofen axetil (medium dose 200 mg, for postoperative analgesia) was also associated with a slightly longer survival but not statistically significant (HR 0.81, 95% CI 0.63-1.03; P = 0.083). Further analysis showed that combined administration of dexamethasone and flurbiprofen axetil had additive effect in prolonging survival (compared to no use of both: adjusted HR 0.57, 95% CI 0.38-0.84, P = 0.005).

The investigators hypothesize that, for patients undergoing surgery for non-small-cell lung cancer, perioperative administration of dexamethasone and flurbiprofen axetil may improve long-term survival. However, evidences from randomized controlled trials are still lacking in this aspect.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 85 years old;
2. Diagnose as non-small-cell lung cancer (stage IA-IIIA);
3. Plan to undergo surgical resection;
4. Provide written informed consents.

Exclusion Criteria:

1. Clinical evidences suggest remote metastasis of the primary cancer; have received radiotherapy, chemotherapy or targeted therapy before surgery; have received previous surgery for lung cancer; diagnosed with other cancer (other than lung cancer) currently or previously;
2. History of therapy with glucocorticoids or immunosuppressants within 1 year, or therapy with non-steroidal anti-inflammatory drugs (NSAIDs) within 1 month;
3. Allergy to glucocorticoids or NSAIDs;
4. Contraindications to dexamethasone or flurbiprofen axetil, such as asthma or hives urticaria induced by aspirin or other NSAIDs; active digestive tract ulcer or bleeding, or history of repeated digestive tract ulcer or bleeding; coagulopathy (platelet count < 50*10^9/L, International Normalized Ratio > 1.4, or activated partial thromboplastin time > 4 seconds above upper limit); current therapy with lomefloxacin, norfloxacin, or enoxacin; severe cardiac dysfunction (New York heart association class 3 or above, or Left Ventricular Ejection Fraction less than 30%) or myocardial infarction within 3 months; liver injury (transaminase higher than 2 times of upper limit); kidney injury (creatinine higher than 1.5 times of upper limit); uncontrolled severe hypertension before surgery (> 180/120 mmHg);
5. ASA physical status class IV or higher;
6. Refuse to use patient-controlled analgesia pump after surgery;
7. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
3-year survival after surgery | From end of surgery until 3 years after surgery.
  Duration of survival within 3 years after surgery.

SECONDARY OUTCOMES:
Survival rates at different times after surgery | At 6 months and 1, 2, 3 years after surgery.
  Survival rates at 6 months and 1, 2, 3 years after surgery.
Duration of recurrence-free survival | From end of surgery until 3 years after surgery.
  Duration of recurrence-free survival within 3 years after surgery
Recurrence-free survival rates at different times after surgery | At 6 months and 1, 2, 3 years after surgery.
  Recurrence-free survival rates at 6 months and 1, 2, 3 years after surgery.
Quality of life (WHOQOL-BREF) at 3 years after surgery | At 3 years after surgery.
  Assessed with World Health Organization Quality of Life Brief Scale (WHOQOL-BREF).
Cognitive function (TICS-m) at 3 years after surgery | At 3 years after surgery.
  Assessed with Telephone Interview for Cognitive Status-modified (TICS-m).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neeman E, Ben-Eliyahu S. Surgery and stress promote cancer metastasis: new outlooks on perioperative mediating mechanisms and immune involvement. Brain Behav Immun. 2013 Mar;30 Suppl(Suppl):S32-40. doi: 10.1016/j.bbi.2012.03.006. Epub 2012 Apr 4. PMID 22504092
- [Background] Ben-David B. Anaesthesia in Cancer Surgery: Can it Affect Cancer Survival? Curr Clin Pharmacol. 2016;11(1):4-20. doi: 10.2174/1574884711666160122093154. PMID 26638975
- [Background] Cassinello F, Prieto I, del Olmo M, Rivas S, Strichartz GR. Cancer surgery: how may anesthesia influence outcome? J Clin Anesth. 2015 May;27(3):262-72. doi: 10.1016/j.jclinane.2015.02.007. Epub 2015 Mar 11. PMID 25769963
- [Background] Bugada D, Bellini V, Fanelli A, Marchesini M, Compagnone C, Baciarello M, Allegri M, Fanelli G. Future Perspectives of ERAS: A Narrative Review on the New Applications of an Established Approach. Surg Res Pract. 2016;2016:3561249. doi: 10.1155/2016/3561249. Epub 2016 Jul 18. PMID 27504486
- [Background] Call TR, Pace NL, Thorup DB, Maxfield D, Chortkoff B, Christensen J, Mulvihill SJ. Factors associated with improved survival after resection of pancreatic adenocarcinoma: a multivariable model. Anesthesiology. 2015 Feb;122(2):317-24. doi: 10.1097/ALN.0000000000000489. PMID 25305092
- [Background] Skevington SM, McCrate FM. Expecting a good quality of life in health: assessing people with diverse diseases and conditions using the WHOQOL-BREF. Health Expect. 2012 Mar;15(1):49-62. doi: 10.1111/j.1369-7625.2010.00650.x. Epub 2011 Jan 31. PMID 21281412